CLINICAL TRIAL: NCT06383754
Title: Clareon Intraocular Lens Stability in Vitrectomy Patients: CLOVE Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Nicholas Fung, Clinical Asst Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Clove
Record Dates: First submitted 2024-03-20; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-03

CONDITIONS: Senile Cataract; Epiretinal Membrane; Vitreous Hemorrhage
MeSH Terms: conditions — Epiretinal Membrane; Vitreous Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients are randomised and masked from the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clareon IOL from Alcon (Experimental): Monofocal artificial lens implanted in the eye following cataract surgery
  Interventions: Device: Clareon
- Tecnis 1 from from Precision Lens (Active Comparator): Monofocal 1 piece IOL implanted in the eye following cataract surgery
  Interventions: Device: Tecnis 1

INTERVENTIONS:
Device: Clareon — Monofocal intraocular lens
  Arms: Clareon IOL from Alcon
Device: Tecnis 1 — Monofocal 1 Piece intraocular lens
  Arms: Tecnis 1 from from Precision Lens

SUMMARY:
This prospective randomized controlled trial will be conducted to investigate Clareon intraocular lens (IOL) stability in vitrectomy patients. The investigator plans to target the patients undergoing cataract surgery. A randomized study will be conducted with 2 arms, one with Clareon IOL versus a second arm using the Tecnis 1 In this non-inferiority study, the investigator will compare Clareon IOL from Alcon with the existing Tecnis 1 IOL from Precision Lens which is the commonly used intraocular lens in combined vitrectomy cases in Hong Kong.

DETAILED DESCRIPTION:
All patients will undergo standard phacoemulsification cataract extraction with Clareon IOL or Tecnis 1 IOL by an experienced cataract surgeon. Followed by vitrectomy to treat either, epiretinal membrane or vitreous hemorrhage.

All patients returned for follow-up visits at 1 week, 1 month, and 6 months after surgery for ophthalmic assessments including:

* Visual acuity measured by Early Treatment of Diabetic Retinopathy Study (ETDRS) chart
* Refraction
* Axial movement and tilt measured by Pentacam (OCULUS Optikgeräte GmbH, Germany) using the Sasaki method. The Scheimpflug image of the horizontal cross-section and the vertical cross-section of the IOL will be selected for measurement. Central ACD will be measured as the distance between the central corneal posterior endothelium to the anterior surface of IOL. The subtraction in ACD between two visits indicated forward or backward axial movement of the IOL.
* Decentration will be measured from the center of the IOL anterior surface to the pupillary axis, which will be perpendicular to the line between the two anterior chamber angles and through the midpoint of the line.
* Tilt will be measured as the angle between the IOL axis and the perpendicular visual axis.
* Any surgical complications and post-op complications will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of senile cataracts and epiretinal membranes or vitreous hemorrhage
* Age between 50 and 80 years.

Exclusion Criteria:

* Diagnosis of vision-impairing diseases including uveitis, glaucoma and corneal pathologies resulting in high astigmatism, severe refractive error (preoperative spherical equivalent of either eye >-6.00D or +5.00D);
* Diagnosis of possible lenses instability including History of ocular trauma, Pseudoexfoliation syndrome; past refractive surgery or other ophthalmic surgery;
* Known Capsular or zonular disorders that might affect the post-operative centration of IOLs, e.g., pseudo-exfoliation syndrome or Marfan syndrome;
* Surgical complications including severe hyphema, iris injury, repeated IOL implantation during surgery, failure to achieve in-the-bag IOL implantation, posterior capsular rupture, usage of tamponade (gas or oil) and corneal sutures.
* Difficulty in obtaining IOL measurements (eg. Small pupil, corneal opacities, patient cooperation)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Position stability of Clareon and Tecnis 1 IOL | 1 week, 1 month and 6 months
  Two arms will compare Intraocular lens stability, which will be measured by it's tilt, measures in degrees from iris plane (0, deg). Tilt will be measured using Pentacam by Sasaki method.

SECONDARY OUTCOMES:
Visual acuity | 1 week, 1 month and 6 months
  Visual acuity will be measured by Early Treatment of Diabetic Retinopathy Study (ETDRS) chart
Refraction | 1 week, 1 month and 6 months
  Refraction will be measured by an autorefractor, and the unit of measurement is Diopter.
Axial movement | 1 week, 1 month and 6 months
  Axial movement will be measured by Pentacam (OCULUS Optikgeräte GmbH, Germany) using the Sasaki method. For axial movement unit of measurement is millimeter.
Decentration | 1 week, 1 month and 6 months
  Decentration will be measured from the center of the IOL anterior surface to the pupillary axis, which will be perpendicular to the line between the two anterior chamber angles and through the midpoint of the line. The unit of measurement for decentration is millimeter.
Compare intra operative and post operative complication | 1 week, 1 month and 6 months
  Any surgical complications and post operative complications will be documented.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Fung, Principal Investigator — The University of Hong Kong
Locations (1):
- Grantham Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
By direct contact to the corresponding author or PI
Supporting Information: Study Protocol, CSR
Time Frame: 5 years after the study ends
Access Criteria: Case by case

REFERENCES:
- [Background] Nagy ZZ, McAlinden C. Femtosecond laser cataract surgery. Eye Vis (Lond). 2015 Jun 30;2:11. doi: 10.1186/s40662-015-0021-7. eCollection 2015. PMID 26605364
- [Background] Korynta J, Bok J, Cendelin J. Changes in refraction induced by change in intraocular lens position. J Refract Corneal Surg. 1994 Sep-Oct;10(5):556-64. PMID 7530106
- [Background] Wang L, Koch DD. Effect of decentration of wavefront-corrected intraocular lenses on the higher-order aberrations of the eye. Arch Ophthalmol. 2005 Sep;123(9):1226-30. doi: 10.1001/archopht.123.9.1226. PMID 16157803
- [Background] Rosales P, Marcos S. Phakometry and lens tilt and decentration using a custom-developed Purkinje imaging apparatus: validation and measurements. J Opt Soc Am A Opt Image Sci Vis. 2006 Mar;23(3):509-20. doi: 10.1364/josaa.23.000509. PMID 16539046
- [Background] de Castro A, Rosales P, Marcos S. Tilt and decentration of intraocular lenses in vivo from Purkinje and Scheimpflug imaging. Validation study. J Cataract Refract Surg. 2007 Mar;33(3):418-29. doi: 10.1016/j.jcrs.2006.10.054. PMID 17321392
- [Background] Dolgin E. The myopia boom. Nature. 2015 Mar 19;519(7543):276-8. doi: 10.1038/519276a. No abstract available. PMID 25788077
- [Background] Schulz KF, Grimes DA. Unequal group sizes in randomised trials: guarding against guessing. Lancet. 2002 Mar 16;359(9310):966-70. doi: 10.1016/S0140-6736(02)08029-7. PMID 11918933
- [Background] Pan CW, Liu H, Sun HP, Xu Y. Increased Difficulties in Managing Stairs in Visually Impaired Older Adults: A Community-Based Survey. PLoS One. 2015 Nov 6;10(11):e0142516. doi: 10.1371/journal.pone.0142516. eCollection 2015. PMID 26545238
- [Background] Lane S, Collins S, Das KK, Maass S, Thatthamla I, Schatz H, Van Noy S, Jain R. Evaluation of intraocular lens mechanical stability. J Cataract Refract Surg. 2019 Apr;45(4):501-506. doi: 10.1016/j.jcrs.2018.10.043. Epub 2019 Jan 25. PMID 30686704